CLINICAL TRIAL: NCT04710537
Title: Comparing AlloDerm and DermACELL in Breast Reconstruction: A Randomized Laterality
Brief Title: Comparing AlloDerm and DermACELL in Breast Reconstruction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: IRB00248878
Record Dates: First submitted 2020-12-29; First posted 2021-01-14 (Actual); Last update posted 2022-08-04 (Actual); Status verified 2022-08

CONDITIONS: Acellular Dermal Matrix in Breast Reconstruction
MeSH Terms: interventions — Alloderm

STUDY DESIGN:
Intervention Model Description: At the time of surgery, the assignment of AlloDerm vs. DermACELL to the patient's left and right breasts will be randomized. The surgical assistant, scrub tech, and circulators can randomly choose which acellular dermal matrix product will be used "first" or "second". The ADM product that will be used first will be placed in either the left or right breast, depending on what breast the surgeon decided to perform the surgery on first. Then, the second breast that is operated on will receive whichever ADM product was not used on the first breast.
Who Masked: Participant, Care Provider
Masking Description: At the time of surgery, the surgeon will be blinded to which acellular dermal matrix product he or she is utilizing in each breast, and the technical steps of the procedure will proceed identically on each side. This can be done through the help of circulators and scrub techs during the surgery, who can randomly prepare either AlloDerm or DermACELL to be placed in either the right or left breast, without informing the surgeon. Other items, like the selection of suture and number of drains placed will be at the discretion of the surgeon but will proceed identically in the two breasts.
  Patients will also be blinded as to what product is in each breast. On the day of surgery, the circulator/operating room assistants will record what product is placed in each breast in the surgery electronic medical note.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AlloDerm (Active Comparator): AlloDerm will be surgically implanted into each participant (either in their left or right breast) at the time of their breast reconstruction surgery. AlloDERM will be placed in the breast opposite to the breast in which DermACELL is placed, so that the patient has AlloDERM in the right breast and DermACELL in the left breast, or vice versa.
  Interventions: Other: AlloDerm
- DermACELL (Active Comparator): DermACELL will be surgically implanted into each participant (either in their left or right breast) at the time of their breast reconstruction surgery. DermACELL will be placed in the breast opposite to the breast in which AlloDERM is placed, so that the patient has AlloDERM in the right breast and DermACELL in the left breast, or vice versa.
  Interventions: Other: DermACELL

INTERVENTIONS:
Other: AlloDerm — Enrolled patients will have one of their breasts reconstructed with AlloDerm at the time of their breast reconstruction surgery.
  Arms: AlloDerm
Other: DermACELL — Enrolled patients will have one of their breasts reconstructed with DermACELL at the time of their breast reconstruction surgery.
  Arms: DermACELL

SUMMARY:
This study will compare 90-day complication rates between breasts reconstructed with tissue expanders and AlloDerm vs. DermACELL, with each patient serving as her own comparator.

DETAILED DESCRIPTION:
The investigators' study aims to determine if there is a significant difference in postoperative outcomes when using DermACELL or AlloDerm, two acellular dermal matrix products, in breast reconstruction. Patients who are undergoing bilateral mastectomies with tissue expanders and acellular dermal matrix (ADM) with one of the investigators' two surgeons, Dr. Steven Davison or Dr. Ximena Pinell, are eligible to be enrolled. Patients' breasts will be randomized to receive either AlloDerm or DermACELL so that each patient had AlloDerm placed in one breast and DermACELL placed in the other on the day of surgery. Then, the following data for each breast will be recorded: time until drain removal, total drain output, time until first expander fill, and occurrences of infection and seroma.

ELIGIBILITY:
Inclusion Criteria:

* Female patients over the age of 18
* May be undergoing either therapeutic or prophylactic mastectomy
* Must be undergoing bilateral mastectomy and breast reconstruction with tissue expanders

Exclusion Criteria:

* Patients who wish to avoid the use of ADM in their reconstruction
* History of radiation of the breast
* Unilateral mastectomies
* Direct to implant breast reconstruction (not utilizing a tissue expander)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Cis-women
Enrollment: 50 (Actual)
Dates: Start 2021-10-21 (Actual); Primary Completion 2022-07-26 (Actual); Study Completion 2022-07-26 (Actual)

PRIMARY OUTCOMES:
Drain time | Up to 90 days
  Number of days between surgical placement of drains and time until drains are removed.
Drain output | Up to 90 days
  Total amount of fluid collected by the drains until their removal (measured in cc).
Incidence of Seroma | Up to 90 days
  Each patient will be evaluated for incidence of seroma in either breast at postoperative visits.
Incidence of Infection | Up to 90 days
  Each patient will be evaluated for incidence of infection in either breast at postoperative visits.

SECONDARY OUTCOMES:
Incidence of Skin necrosis | Up to 90 days
  Each patient will be evaluated for skin necrosis of either breast at postoperative visits.
Incidence of Hematoma | Up to 90 days
  Each patient will be evaluated for incidence of hematoma in either breast at postoperative visits.
Incidence of Device Explantation | Up to 90 days
  If patients require device explantation in one breast due to complications (e.g. infection).

CONTACTS AND LOCATIONS:
Overall Officials: Steven P Davison, MD, Principal Investigator — Sibley Memorial Hospital
Locations (2):
- United States (2):
  - DAVinci Plastic Surgery, Washington D.C., District of Columbia
  - Sibley Memorial Hospital, Washington D.C., District of Columbia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zenn MR, Salzberg CA. A Direct Comparison of Alloderm-Ready to Use (RTU) and DermACELL in Immediate Breast Implant Reconstruction. Eplasty. 2016 Aug 11;16:e23. eCollection 2016. PMID 27602176
- [Background] Pittman TA, Fan KL, Knapp A, Frantz S, Spear SL. Comparison of Different Acellular Dermal Matrices in Breast Reconstruction: The 50/50 Study. Plast Reconstr Surg. 2017 Mar;139(3):521-528. doi: 10.1097/PRS.0000000000003048. PMID 28234811
- [Background] Steiner CA, Weiss AJ, Barrett ML, Fingar KR, Davis PH. Trends in Bilateral and Unilateral Mastectomies in Hospital Inpatient and Ambulatory Settings, 2005-2013. 2016 Feb [updated 2016 Mar]. In: Healthcare Cost and Utilization Project (HCUP) Statistical Briefs [Internet]. Rockville (MD): Agency for Healthcare Research and Quality (US); 2006 Feb-. Statistical Brief #201. Available from http://www.ncbi.nlm.nih.gov/books/NBK367629/ PMID 27253008